CLINICAL TRIAL: NCT05122884
Title: Effect of Milrinone Versus Placebo on Hemodynamics in Patients With Septic Shock; Randomized Control Trial
Brief Title: Milrinone Versus Placebo in Patients With Septic Shock
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SI 111/2021
Record Dates: First submitted 2021-09-23; First posted 2021-11-17 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Septic Shock; Cardiac Output
Keywords: Milrinone; Septic shock; Cardiac output; Poor tissue perfusion
MeSH Terms: conditions — Shock, Septic | interventions — Milrinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacist who does not involve in patient enrollment nor treatment will prepared milrinone or placebo in the identical container, before the study drug will be given to patients, according to their treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Milrinone group (Experimental): The pharmacist prepares milrinone 20 mg with normal saline solution (NSS) 100 ml then starts dose 0.5 mg/kg/min for up to 12 hours. The doctor performs Echocardiogram before start Milrinone, during infusion, and after 12 hours from stop Milrinone. Other medications or interventions were used or not used depending on own doctor.
  Interventions: Drug: Milrinone
- Placebo group (Placebo Comparator): The pharmacist uses 100 ml of NSS, packed out in the same format, dose, and administration of the drug were exactly the same as in the milrinone group. The doctor performs Echocardiogram same time as the milrinone group
  Interventions: Drug: Milrinone

INTERVENTIONS:
Drug: Milrinone — Prepare milrinone 20 mg with NSS 100 ml then starts dose 0.5 mg/kg/min for up to 12 hours.
  Other Names: Primacor

SUMMARY:
Sepsis is one of the most serious healthcare problems, worldwide, and financial burdens.

The overall mortality of severe sepsis/septic shock was 44.5-52.6%. A common cause of death is refractory shock and multi-organ failure. Myocardial dysfunction is a relatively common complication of septic shock. This causes a decrease in the amount of cardiac output, resulting in insufficient blood supply to the organ and multi-organ failure and lead to death Early goal-directed therapy began to use dobutamine in patients with septic shock Sepsis Survival Campaign Guideline 2016 recommended drug is dobutamine and an alternative drug is milrinone in septic shock patients with clinical signs of poor tissue perfusion.

DETAILED DESCRIPTION:
According to several studies, the use of dobutamine increases the amount of cardiac output but it has also been reported to increase mortality rates too. There are few studies of milrinone in patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Diagnosis Septic Shock from the definition of SEPSIS III in intensive care unit at Siriraj hospital and Hat-Yai hospital
* Receive fluid resuscitation at least 30 ml/kg and/or Vasopressor until mean arterial pressure ≥ 65 mmHg
* Persistence lactate >2mmol/L at 6th hour after resuscitation
* Urine output < 0.5 ml/kg at 6th hour after resuscitation
* Left ventricular ejection fraction (LVEF) < 40 %

Exclusion Criteria:

* Chronic kidney disease stage 5 and denied renal replacement therapy
* Life-threatening tachyarrhythmia before enrolled e.g. Ventricular tachycardia, Ventricular fibrillation
* Patient sign do-not-resuscitation and terminally ill

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The change of cardiac output from baseline (before study drug administration) to 6 hours (during study administration) | upto 24 hours
  by echocardiogram or Pulse contour analysis or Thermodilution technique from pulmonary artery catheter

SECONDARY OUTCOMES:
Intensive care unit (ICU) mortality | upto 120 days
  Proportion of participant who die during ICU admission
Hospital mortality | upto 120 days
  Proportion of participant who die during hospital admission
28-day mortality | upto 28 days
  Proportion of participant who die during 28 days after enrollment
Dose of vasopressor after intervention | upto 7 days
  present as vasopressor equivalent dose compare before and after intervention, and percent of decrease
Lactate clearance | upto 7 days
  lactate level after and before intervention and percent clearance
Mechanical ventilator free day | upto 28 days
  day of the patient does not use mechanical ventilator during admission
Extracorporeal membrane oxygenation (ECMO) or Renal replacement therapy (RRT) | upto 28 days
  incident of initial ECMO or RRT
Incident of tachyarrhythmia | upto 28 days
  Incident of ventricular tachycardia, ventricular fibrillation, Atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Surat Tongyoo, Principal Investigator — Mahidol University
Locations (2):
- Thailand (2):
  - Hat Yai Hospital, Hat Yai, Changwat Songkhla
  - Department of Medicine, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
Anonymous identification data will be prepared per request, after study publication 6 months.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 6 months post study publication
Access Criteria: Request to principal investigation, after protocal approval from ethical committee.

REFERENCES:
- [Derived] Tongyoo S, Chobngam S, Yolsiriwat N, Jiranakorn C. Effects of adjunctive milrinone versus placebo on hemodynamics in patients with septic shock: a randomized controlled trial. Ann Med. 2025 Dec;57(1):2484464. doi: 10.1080/07853890.2025.2484464. Epub 2025 Mar 26. PMID 40138463